CLINICAL TRIAL: NCT05944120
Title: Decreasing On-Shift Stress With a Crisis Intervention Cart
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 006.NUR.2022.A
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Decreasing On-Shift Stress With a Crisis Intervention Cart

STUDY DESIGN:
Intervention Model Description: As noted in the background, resiliency-building activities appear to have a positive relationship with managing stress in the workplace. Additionally, offering a variety of strategies is anticipated to increase the sample size and encourage continued use of the strategies over time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Crisis Intervention Cart (Experimental): To determine if a Crisis Intervention Cart filled with evidence-based stress-reducing interventions does reduce stress experienced during a shift.
  Interventions: Combination Product: Aromatherapy patches

INTERVENTIONS:
Combination Product: Aromatherapy patches — This study anticipates that Staff-reported stress levels will decrease when nurses use strategies from the Crisis Intervention Cart while at work.
  Other Names: Crisis Intervention Cart deployment.

SUMMARY:
This Intervention study anticipates that 100 nurses, patient care technicians and unit secretaries in the acute care setting at four Methodist Health System facilities will provide surveys to participants who had interventions

DETAILED DESCRIPTION:
Once the intervention has been used, the participants will complete a survey in order to determine if stress levels are decreasing. Initial data collection will be over the course of two months ( April 1, 2022 through June 1, 2022) and participation will vary based upon staffing and the set criteria for Crisis Intervention Cart deployment.

ELIGIBILITY:
Inclusion Criteria:

* Part of MHS (i.e., MCMC, MMMC, MRMC, MDMC, MLMC, MSMC)
* The hospital has at least one Crisis Intervention Cart study clinical site investigator on-staff
* Hold license as a Registered Nurse OR
* Hold position as a patient care technician or unit secretary
* Must be able to read English
* Provide direct patient care or hold a unit-based leadership position (i.e., Nursing Clinical Coordinator, Nurse Manager, Clinical Team Lead)
* Full-time, part-time, or PRN employee

Exclusion Criteria:

* Hospitals and clinical units will be excluded if they are outside MHS
* Participants will be excluded if they at Director-level or above

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Crisis Intervention Cart | Period of 2 months
  The Effect of Crisis Intervention Cart filled with evidence-based stress-reducing interventions on reducing stress experienced during a shift using surveys. A 10-point Likert scale will be used with 1 being the lowest and 10 being the highest on the scale with 10 having highest level of self-perceived stress.

SECONDARY OUTCOMES:
Type of intervention/strategy used | Period of 2 months
  The Effect of Crisis Intervention Cart filled with evidence-based stress-reducing interventions on reducing stress experienced during a shift using surveys. A 10-point Likert scale will be used with 1 being the lowest and 10 being the highest on the scale with 10 having the highest level of self-perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Cheyenne Ruby, DNP, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Badu E, O'Brien AP, Mitchell R, Rubin M, James C, McNeil K, Nguyen K, Giles M. Workplace stress and resilience in the Australian nursing workforce: A comprehensive integrative review. Int J Ment Health Nurs. 2020 Feb;29(1):5-34. doi: 10.1111/inm.12662. PMID 31917519
- [Background] Labrague LJ, de Los Santos JAA. Resilience as a mediator between compassion fatigue, nurses' work outcomes, and quality of care during the COVID-19 pandemic. Appl Nurs Res. 2021 Oct;61:151476. doi: 10.1016/j.apnr.2021.151476. Epub 2021 Jul 7. PMID 34544570
- [Background] Mintz-Binder R, Andersen S, Sweatt L, Song H. Exploring Strategies to Build Resiliency in Nurses During Work Hours. J Nurs Adm. 2021 Apr 1;51(4):185-191. doi: 10.1097/NNA.0000000000000996. PMID 33734177
- [Background] Haddad LM, Annamaraju P, Toney-Butler TJ. Nursing Shortage. 2023 Feb 13. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK493175/ PMID 29630227
- [Background] Manomenidis G, Panagopoulou E, Montgomery A. Resilience in nursing: The role of internal and external factors. J Nurs Manag. 2019 Jan;27(1):172-178. doi: 10.1111/jonm.12662. Epub 2018 Jul 31. PMID 30066352
- [Background] Restrepo J, Lemos M. Addressing psychosocial work-related stress interventions: A systematic review. Work. 2021;70(1):53-62. doi: 10.3233/WOR-213577. PMID 34511476
- [Background] Velana M, Rinkenauer G. Individual-Level Interventions for Decreasing Job-Related Stress and Enhancing Coping Strategies Among Nurses: A Systematic Review. Front Psychol. 2021 Jul 19;12:708696. doi: 10.3389/fpsyg.2021.708696. eCollection 2021. PMID 34349711